CLINICAL TRIAL: NCT01543243
Title: Application of Whole-body Vibration With Stochastic Resonance in Frail Elderly: The Effects on Postural Control: a Pilot Study
Brief Title: Application of Whole-body Vibration With Stochastic Resonance in Frail Elderly: The Effects on Postural Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Goethe University (Other); Maastricht University Medical Center (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Slavko Rogan, cand. PhD, PTMsc, PT MSc, Bern University of Applied Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PhD pilot study 2
Record Dates: First submitted 2011-09-26; First posted 2012-03-02 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Equilibration Disorder, Vestibular Nerve
Keywords: postural balance; strength

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1: immediate effects: T0, Stochastic resonance whole-body vibration A intervention, immediate T1 (one minute after Stochastic resonance whole-body vibration B intervention), 7 days wash-out period; T2, Stochastic resonance whole-body vibration intervention, immediate T3 (one minute after Stochastic resonance whole-body vibration intervention)
  long term effect: T4, Stochastic resonance whole-body vibration A intervention over four weeks, three time a week;T5, 16 days wash-out period; T6, Stochastic resonance whole-body vibration B intervention over four weeks, three times week, T7
  Interventions: Device: Stochastic resonance whole-body vibration A; Device: Stochastic resonance whole-body vibration B
- Group 2 (Experimental): Group 2: immediate effect: T0, Stochastic resonance whole-body vibration B intervention, immediate T1 (one minute after intervention), 7 days wash-out period; T2, Stochastic resonance whole-body vibration A intervention, immediate T3 (one minute after intervention)
  Long term effect: T4, Stochastic resonance whole-body vibration B intervention over four weeks, three time a week;T5, 16 days wash-out period;T6, Stochastic resonance whole-body vibration A intervention over four weeks, three times week, T7
  Interventions: Device: Stochastic resonance whole-body vibration A; Device: Stochastic resonance whole-body vibration B

INTERVENTIONS:
Device: Stochastic resonance whole-body vibration A — Immediate effects (one minute after intervention): over 5 sets with 6 Hz, Noise 4 and than 1 Hz, Noise 1.
  Long term effect: over four weeks, three times a week with 6 Hz, Noise 4 and than over four weeks three times a week with 1 Hz, Noise 1.
  Other Names: SRT Zeptor® med plus Noise
Device: Stochastic resonance whole-body vibration B — Immediate effects (one minute after intervention): over 5 sets with 1 Hz, Noise 1 and than 6 Hz, Noise 4.
  Long term effect: over four weeks, three times a week with 1 Hz, Noise 1 and than four weeks three times a week with 6 Hz, Noise 4.
  Other Names: SRT Zeptor® med plus Noise

SUMMARY:
This study aims to examine

1. the feasibility
2. immediately
3. long term effects on postural control and strength of mechanical SR-WBV intervention in a frail elderly population.

DETAILED DESCRIPTION:
This study is based on the guideline of falls management exercise programs (FaME) designed exercise from Skelton and Dinan.

The FAME program is structured so that four biocybernetic pillars are embedded in the three successive stages of training.

The biocybernetic pillars:

1. improving the balance
2. improvement in functional capacity
3. improvement in bone density and muscle mass Overthrowing 4) improving the security (reducing anxiety).

The training phase should reach the following goals:

1. Skilling up: with the aim of improving improve neuromuscular control, postural control and strengthening of large muscle groups of the lower extremity.
2. Training Gain: with the aim to improve functional abilities.
3. Maintaining the Gains: with the goal of muscle mass and bone density and introduce them to build complex multi-sensory exercises.

We started the FaME program with assistance from the pilot study, "Effects of stochastic resonance therapy on postural control in the elderly population" (KEK Bern: No.228/09, Trial Registry: NCT01045746). It was found that a whole-body vibration with stochastic resonance (SR-WBV) enables that strength, coordination, and balance training while standing, in the exercise training gain phase is possible.

For this reason, this study will examine the feasibility and the immediately and long term effects of SR-WBV with 6 Hz, Noise 4 on postural control and strength in frail elderly.

ELIGIBILITY:
Inclusion Criteria:

* RAI (Resident Assessment Instrument) >0
* live in canton Bern
* in terms of training load be resistant.

Exclusion Criteria:

* acut joint disease, acut thrombosis, acute fractures, acute infections, acute tissue damage, or acute surgical scars
* seniors with prosthesis.
* alcoholic
* acute joint disease, activated osteoarthritis, rheumatoid arthritis, acute lower limb
* acute inflammation or infection tumors
* fresh surgical wounds
* severe migraine
* epilepsy
* acute severe pain

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Dynamic body balance | effects after 4 weeks
  The Expanded Timed Get Up-and-Go (ETGUG) will be used for measuring dynamic body balance. At 2, 8 and 10 meters along the walkway, markers were set, allowing to the measurement the change of the split times.

SECONDARY OUTCOMES:
static body balance | immediate effects following one minute after a session of SR-WBV
  Semi-tandem stand (STS): Anterior-posterior (AP) and medial-lateral (ML) sway on a force plate during the STS will be measured.
static body balance | effects after 4 weeks
  Semi-tandem stand (STS): Anterior-posterior (AP) and medial-lateral (ML) sway on a force plate during the STS will be measured.
dynamic body balance | immediate effects following one minute after a session of SR-WBV
  The Expanded Timed Get Up-and-Go (ETGUG) will be used for measuring dynamic body balance. At 2, 8 and 10 meters along the walkway, markers were set, allowing to the measurement the change of the split times.
dynamic body balance | effects after 4 weeks
  The Expanded Timed Get Up-and-Go (ETGUG) will be used for measuring dynamic body balance. At 2, 8 and 10 meters along the walkway, markers were set, allowing to the measurement the change of the split times
Lower extremity performance | immediate effects following one minute after a session of SR-WBV
  Short physical performance battery (SPBB):The SPPB combines the results of balance tests (semi-tandem stand, side-by-side stand,full tandem stand), gait speed, and chair rise tests.
Lower extermity performance | effects after 4 weeks
  Short physical performance battery (SPBB):The SPPB combines the results of balance tests (semi-tandem stand, side-by-side stand,full tandem stand), gait speed, and chair rise tests.
strength | immediate effects following one minute after a session of SR-WBV
  Muscle strength: It will be evaluated by five-sit-to-stand test and isometric rate of forcedevelopment and isometric Maximum Voluntary Contraction (MCV).
strength | effects after 4 weeks
  Muscle strength: It will be evaluated by five-sit-to-stand test and isometric rate of forcedevelopment and isometric Maximum Voluntary Contraction (MCV).

CONTACTS AND LOCATIONS:
Overall Officials: Slavko Rogan, MSc, Study Chair — Bern University of Applied Science, Department Health; Lorenz Radlinger, PhD, Principal Investigator — Bern University of Applied Science, Department Health; Dietmar Schmidtbleicher, PhD, Prof., Study Director — Johann Wolfgang Goethe University Frankfurt am Main, Department Sport Science; Rob de Bie, PhD, Prof., Study Director — University Maastricht, Department Epidemiology; Eling D de Bruin, PhD, Prof., Study Director — Swiss Federal Institute of Technology Zurich, Department Human Movement Science
Locations (1):
- Bern University of Applied Science, Department Health, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Result] Rogan S, Schmidtbleicher D, Radlinger L. Immediate effects after stochastic resonance whole-body vibration on physical performance on frail elderly for skilling-up training: a blind cross-over randomised pilot study. Aging Clin Exp Res. 2014 Oct;26(5):519-27. doi: 10.1007/s40520-014-0212-4. Epub 2014 Apr 4. PMID 24700493
- [Result] Rogan S, Radlinger L, Schmidtbleicher D, de Bie RA, de Bruin ED. Preliminary inconclusive results of a randomised double blinded cross-over pilot trial in long-term-care dwelling elderly assessing the feasibility of stochastic resonance whole-body vibration. Eur Rev Aging Phys Act. 2015 Oct 9;12:5. doi: 10.1186/s11556-015-0150-y. eCollection 2015. PMID 26865869